CLINICAL TRIAL: NCT02425839
Title: Assessment of Correlation Between Changes of Shear Wave Elastography and Surface Electromyogram of the Masseter, in Rest and Maximal Voluntary Contraction
Brief Title: Assessment of Correlation Between Changes of Shear Wave Elastography and Surface Electromyogram of the Masseter
Acronym: EVEREST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 1408203; 2015-A00073-46 (Other: ANSM)
Record Dates: First submitted 2015-04-09; First posted 2015-04-24 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Masseter Muscle Spasm
Keywords: shear wave elastography; surface electromyogram; masseter
MeSH Terms: conditions — Trismus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental group (Experimental): * ultrasound exam by Supersonic Shear Imaging® technique
  * EMG examination by electromyograph Keypoint system.
  Interventions: Device: Ultrasound exam by Supersonic Shear Imaging® technique; Device: EMG examination by electromyograph Keypoint system

INTERVENTIONS:
Device: Ultrasound exam by Supersonic Shear Imaging® technique — Each of the two observers performs twice ultrasound examination and measures of the masseter thickness and its elastic modulus, at rest and maximal voluntary contraction.
Device: EMG examination by electromyograph Keypoint system — Experimented neurologist performs EMG examination.

SUMMARY:
Diagnoses and follow up of muscles diseases lack imaging. Severity assessment of masticatory dysfunction and follow up of treatment effectiveness is currently based only on clinical features. Supersonic ShearWave Imaging® is a new, non-invasive, non-irradiating and dynamic imaging technique that uses ultrasound and allows shear wave elastic modulus in a muscle in order to study its viscoelastic properties.

In this study, the investigators study the correlation between changes of shear wave elastography modulus and surface electromyogram features of the masseters between rest and maximal voluntary contraction.

ELIGIBILITY:
Inclusion Criteria:

* People with social security.
* People aged 20 to 40 years, of both sexes.
* People that gave and signed consent to participate in the study.

Exclusion Criteria:

* Any concomitant muscle disease (myopathy, myositis…)
* Botulinum toxin injections in the masseter in the last 3 months preceding the study.
* Any treatment that induces muscular effect (baclofen, benzodiazepine)
* Bruxism or any masticatory apparatus disease
* Any surgery of the masticatory apparatus

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Elastic modulus using Supersonic Shear Imaging® technique on superficial and deep masseter parts at rest and maximal voluntary contraction. | Day 1 (inclusion day)

SECONDARY OUTCOMES:
Thickness of the whole masseter mesured by Supersonic Shear Imaging® technique | Day 1 (inclusion day)
Thickness of the masseter superficial part mesured by Supersonic Shear Imaging® technique | Day 1 (inclusion day)
Thickness of the masseter deep part mesured by Supersonic Shear Imaging® technique | Day 1 (inclusion day)

CONTACTS AND LOCATIONS:
Overall Officials: Claire BOUTET, MD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France